CLINICAL TRIAL: NCT06919614
Title: Improving PrEP Outcomes Among Pregnant Women in Botswana With an Integrated STI Testing and PrEP Delivery Model
Brief Title: STI Testing to Enhance PrEP Use in Pregnancy
Acronym: STEP-UP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Botswana Harvard AIDS Institute Partnership (Other)
Collaborators: University of Washington (Other); University of Botswana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BHP180
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: PrEP Adherence; Sexually Transmitted Infections (STIs); Pregnancy
Keywords: Pregancy; PrEP; HIV; STIs; Chlamydia; Gonorrhoea; Gonorrhea; Trichomonas; Dapivirine; Truvada; Oral PrEP
MeSH Terms: conditions — Sexually Transmitted Diseases; Chlamydia Infections; Gonorrhea; Trichomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Participants randomized to the intervention arm will be offered Xpert® CT/NG and TV testing and treatment (in addition to syndromic STI assessment) at three time points (enrolment, at the 32 weeks' gestation visit and 9-month post-delivery visit) or two time points for participants enrolled in their third trimester. If a client accepts Xpert® testing, they will be instructed by the study clinician/research assistant on how to self-collect a vaginal swab.
  Interventions: Diagnostic Test: Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis testing
- Standard-of-care arm (No Intervention): Participants in the standard-of-care arm will receive syndromic STI assessment per Botswana national guidelines. They will be offered Xpert® CT/NG and TV testing at the 9-month post-delivery visit only.

INTERVENTIONS:
Diagnostic Test: Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis testing — Xpert® CT/NG and TV testing
  Arms: Intervention arm

SUMMARY:
The investigators are conducting a study in Botswana to see if offering STI testing along with expanded HIV prevention options (PrEP) helps more pregnant women start and continue using PrEP during and after pregnancy. Pregnant women (n=600) seeking antenatal care in Botswana will be enrolled and randomly assigned to receive the standard of care (standard STI assessment with no STI testing) versus STI testing for Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis during pregnancy and postpartum. The investigators' hypothesis is that providing STI testing alongside PrEP offer will encourage more women to start and continue using PrEP.

DETAILED DESCRIPTION:
The investigators are conducting a 2-arm 1:1 randomized trial to compare PrEP delivery with co-offer of STI testing for Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis (using Xpert CT/NG and TV assays) vs. standard-of-care (SOC, syndromic management) among pregnant women without HIV (n=600) in Botswana. Antenatal care clients will be offered PrEP (self-select oral pills or DPV-VR).

Participants will be followed up to 9 months postpartum. Women will be able to switch PrEP methods and start, stop, or restart PrEP at any time.

Primary outcomes are the proportion of clients who initiate PrEP, persist with use at 9 months postpartum, and adhere (quantified by hair drug levels). Secondary outcomes are PrEP choice (pills vs. DPV-VR), STI rates, and birth outcomes by randomization arm. Exploratory outcomes are HIV incidence, quality of care, adherence cofactors, and antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and seeking antenatal care
* Self-identifying as a cis-gender woman
* Living without HIV
* Not currently using PrEP
* Planning to remain in the city/town of enrolment until 9 months post-delivery.
* Planning to receive antenatal and postnatal care in the city/town of enrolment.
* Willing and able to provide informed consent

Exclusion Criteria:

* Male gender
* Not pregnant
* Living with HIV
* Currently using PrEP
* Not planning to remain in the city/town of enrolment until 9 months post-delivery
* Not planning to receive antenatal and postnatal care in the city/town to enrolment
* Not able or willing to provide informed consent for participation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation among pregnant women seeking antenatal care | Enrolment to 1 month post enrolment
  PrEP initiation among pregnant women seeking antenatal care defined as accepting either daily oral PrEP pills or the DPV-VR when offered at enrolment and evidence of self-reported use at 1-month.
PrEP persistence | Enrolment to 9 months postpartum
  Evidence of PrEP persistence at 9 months postpartum among women who initiated PrEP.
PrEP adherence | Enrolment to 9 months postpartum
  PrEP adherence defined as either TFV or DPV hair levels (depending on PrEP method) at 9 months postpartum.

SECONDARY OUTCOMES:
PrEP Choice | Enrolment to 9 months postpartum
  Secondary outcomes are PrEP choice (pills vs. DPV-VR)
STI rates | Enrolment to 9 months postpartum
  Prevalence of chlamydia, gonorrhoea and trichomonas at enrolment, third trimester and 9 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- DHMT Clinics, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No